CLINICAL TRIAL: NCT01126333
Title: Long-term Follow-up of Sirolimus-based Therapy Versus Continued Tacrolimus-based Therapy in Renal Allograft Recipients.
Brief Title: Long-term Follow-up of Spare the Nephron (STN) Patients
Acronym: STN
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Matthew R Weir, PI, University of Maryland, Baltimore
Other Study IDs: HP-00042739
Record Dates: First submitted 2010-05-17; First posted 2010-05-19 (Estimated); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Kidney Transplant
Keywords: Nephrotoxicity, Kidney Transplantation, Graft Survival; Kidney transplant survival.

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Long term Sirolimus or Tacrolimus: Ths study cohort will consist of participants who successfully completed two years of the original Spare the Nephron (STN) study, a two year prospective multi-center study where participants were assigned to receive either center-specific CNI regimen (assigned at the time of transplantation) or were switched to replace the CNI with Sirolimus therapy.
  In this current long-term follow-up study, we will approach patients who previously enrolled in the STN study and offer them the opportunity to enroll to be followed-up for another 3 years. There will be no change in immunosuppression unless clinically indicated. The majority of effort is standard care with every 6 month follow-up appointments.Participants will be required to consent to participate in the three year extension study.

SUMMARY:
Allograft nephropathy is the most common cause of allograft failure following kidney transplantation. Among putative etiologies, cumulative exposure to calcineurin inhibitors may be one of the important progression factors.

"Spare the Nephron"(STN) is a unique study. Patients were randomized to either continue center-specific Calcinerium Inhibitor (CNI) therapy or have CNI replaced with sirolimus within the first six months after transplantation. Approximately 305 patients were enrolled in the study. More than 230 patients finished 2 years of follow-up. There was better patient and graft survival in those converted to sirolimus. There was also a 10% improvement in the kidney function of those who were converted. In this cohort, we wish to explore the durability of this improvement.

DETAILED DESCRIPTION:
In this extension study we will be extending our clinical observation of the STN patients from two to five years. It is expected that a Calcinerium Inhibitor (CNI) sparing regimen will be associated with better preservation of kidney function and fewer cardiovascular events.

STN is a prospective multi-center study that has completed enrollment of 305 first time recipients of kidney allografts from 27 centers. The enrollees were randomly assigned either to continue the center-specific CNI regimen (assigned at the time of transplantation) or were switched to replace the CNI with sirolimus therapy. Either CNI or sirolimus are being used in combination with CellCept therapy with or without the use of maintenance steroids, based on individual center preferences. Induction therapy was also center-specific.

In the present long-term follow-up study we will approach patients previously enrolled in the STN study and offer them the opportunity to enroll to be followed for another 3 years. There will be no changes in immunosuppression unless clinically indicated. The majority of the effort is standard care with every 6 month follow-up appointments.They will be required to be consented to participate in the three year extension study.

Research procedures:

The only inclusion criteria is willingness to sign the consent form for the extension study, after successful completion of the two year STN study.

Study entry is defined as the point at which they sign the consent form, and agree to participate in the study extension.All patients will be followed for 3 years from their initial screening visit. There will be 7 visits during the study period. All procedures will be standard care for long-term transplant follow-up, with no changes in immunosuppression unless clinically indicated. The only exception to standard of care is obtaining a 24 hour urine for protein and creatinine clearance every 6 months during the follow-up.

Visit 1 (Study entry) 1. Review of inclusion/exclusion criteria 2. Medical history, recipient's age, gender and race 3. Complete transplant information i. date of transplant ii. tissue and ABO typing iii. B-Cell cross match, PRA iv. Patient/donor EBV and CMV serology

The patients will stay on the same immunosuppression as they were receiving in the STN study, unless medications were changed due to medical reasons. They will be routinely monitored as per center practice.

The drugs are given as standard of care and the extension of this study does not alter the participants' medication regimen.

The following laboratory evaluations are typically performed at each visit.

1. Tacrolimus / sirolimus trough concentration. Immunosuppressive regimen will be reviewed and changed or adjusted as necessary.
2. CBC with differential
3. Chemistry panel: glucose, Na, K, Cl, CO2, Ca, P, Mg, blood urea nitrogen (BUN), albumin and total protein, AST, ALT, bilirubin (total), alkaline phosphatase and serum creatinine 4 Estimated GFR from blood and urine data.

5. Fasting lipid profile: total cholesterol, LDL, HDL, HDL/LDL ratio, triglycerides

The following clinical assessments will also be performed and recorded in each visit: 1. Vital signs 2. Weight measurements 3. Concomitant medications 4. Adverse events 5. Opportunistic infections 6. Malignancies 7. Clinical evaluation of signs or symptoms of rejection

Number of patients with adverse events will be summarized by body system and each adverse event. Incidence of adverse events will also be summarized by severity and relationship to study medication. Any serious adverse events or deaths will be summarized separately. patient death, graft loss, the need to be withdrawn from the original assigned calcineurin inhibitor therapy patients who return to dialysis for 6 or more consecutive weeks, patients who experience adverse events that lead to premature withdrawal or loss to follow-up. Patients will be followed until the end of the study in all cases. All failed patients will be followed until the end of the last follow up visit (36 months) unless consent is withdrawn. The proportion of patients experiencing any opportunistic infections will be summarized up to 6, 12, 24 ,and 36 months after randomization.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female post-transplant patients who were in the Spare-the-nephron study.
2. Patients capable of understanding the purpose and risks of the study, who can give written informed consent and who are willing to participate in and comply with the study.
3. Women of child bearing potential must not be pregnant or breast-feeding.
4. Women of child bearing age must use two reliable forms of contraception simultaneously, unless they are status post bilateral tubal ligation, bilateral oophorectomy or hysterectomy. Effective contraception must be used before beginning of study drug therapy, for duration of study and for 12 weeks following the completion of study.
5. Must pass the evaluation to sign informed consent form.

Exclusion Criteria:

1. Male or female post-transplant patients who were enrolled in the Spare-the-nephron study, however dropped out during the study period.
2. Inability to pass the Evaluation to Sign Consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients who were previously enrolled in the Spare-the-nephron study.
Sampling Method: Non-Probability Sample
Enrollment: 128 (Actual)
Dates: Start 2010-06; Primary Completion 2014-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
To compare between treatment groups, change in renal function as measured by 24 hour creatinine clearance and estimated GFR. | Every 6 months for 3 years.

SECONDARY OUTCOMES:
Graft and patient survival. | Every 6 months for 3 years.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew R Weir, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland Medicine, Division of Adult Nephrology, Baltimore, Maryland, United States